CLINICAL TRIAL: NCT03660995
Title: Better Understanding Slow Language Impairment: Cognitive and Genetic Mechanisms
Brief Title: Better Understanding Slow Language Impairment
Acronym: SLI:COGGEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO18001
Record Dates: First submitted 2018-01-04; First posted 2018-09-07 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Slow Language Impairment
Keywords: Slow language impairment; semantic; pragmatic; procedural learning; genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLI children (Experimental)
  Interventions: Behavioral: Evaluation of language skills and procedural learning of children with SLI and their controls. DNA sampling.
- Control children (Active Comparator)
  Interventions: Behavioral: Evaluation of language skills and procedural learning of children with SLI and their controls. DNA sampling.

INTERVENTIONS:
Behavioral: Evaluation of language skills and procedural learning of children with SLI and their controls. DNA sampling. — Behavioral evaluation of language skills at the formal, semantic and pragmatic levels and of procedural learning for each child with SLI and each control child.
  DNA sampling for each child.

SUMMARY:
This study was designed to examine the development of children aged 6 to 10 with slow language impairment (SLI). The aim was threefold: (1) to investigate language skills of children with SLI at different levels - formal, semantic, pragmatic- in comparison with those of control children; (2) to test a procedural deficit hypothesis: abnormal development in the procedural memory system could account for some language deficits; (3) to make genotype-phenotype comparisons, focusing on the different levels of language development and on procedural skills. The main hypothesis is that genetic mutations, contingently epistatique, will lead to procedural learning deficit, which will have a negative impact on language skills at the formal level and consequently on semantic and pragmatic levels.

DETAILED DESCRIPTION:
To test the main hypothesis, 60 SLI children and 100 controls children will be included on the protocol. Due to the lack of specific standardized tests, the diagnostic of specific language-impaired French children is a challenge. Thus, both a battery of standardized and non-standardized language tests (assessing the different levels: formal, semantic and pragmatic) will be administered to children to establish a profile of weaknesses for each child with SLI and to examine the relationships between SLI and procedural learning. DNA sampling will be conducted on each child, SLI and control, to allow subsequently the molecular analyses in order to run the association comparisons between behavioral data and genetic profiles.

The protocol includes as verbal standardized tests: the Echelle "Vocabulaire en Images Peabody" (EVIP;), the "Epreuve de COmpre´hension Syntaxico-SEmantique" (ECOSSE), two specific subtests (lexicon and grammar) of the "Evaluation du Langage Oral" (ELO;), and as non-standardized tests: a semantic inference task (drawing the meaning of new words from the context, and the meaning of predicative metaphors), and a pragmatic inference task (understanding of indirect requests, on speakers' intention meaning and on irony). The procedural learning skills will be assessed thanks to a serial reaction task, specifically adapted for children).

The complete sequencing of FoXP2 gene, as well as the genotyping of the 44 single nucleotide polymorphisms (SNPs), located in the risk haplotypes identified in ATP2C2, CMIP, CNTNAP2 genes and in the KIAA0319/TTRAP/THEM2 locus, will be conducted.

ELIGIBILITY:
Inclusion Criteria:

For SLI group, the inclusion criteria are:

* To present a slow language impairment
* To speak French

For control group, the inclusion criteria are:

* Being at elementary French school
* Speak French

Exclusion Criteria:

* Child with a neuro-motrice pathology or psychopathology
* Child with a neurological medication
* Child who have a score inferior to percentile 20 on the "Coloured Progressive Matrices" (Raven, 1998)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2019-06-29 (Actual); Primary Completion 2022-05-29 (Estimated); Study Completion 2023-05-29 (Estimated)

PRIMARY OUTCOMES:
Language development | Day 0
  Assessment using :
  * For each of the following tasks, the number of correct answers of children at the questions is collected. These scores can be aggregated (addition).Echelle "Vocabulaire en Images Peabody" (EVIP; Dunn, The´riault-Whalen, & Dunn, 1993). Scale range: 0-170.
  * the "Epreuve de COmpréhension Syntaxico-SEmantique" (ECOSSE; Lecocq, 1996) task. Scale range: 0-92. ,
  * two specific subtests (lexicon and grammar) of the "Evaluation du Langage Oral" (ELO; Khomsi, 2001). Scale range: 0-57, respectively 32 (Lexicon subtest) and 25 'grammar subtest)
  * non-standardized tests: a semantic inference task (drawing the meaning of new words from the context, and the meaning of predicative metaphors), and a pragmatic inference task (understanding of indirect requests, on speakers' intention meaning and on irony). Scale range: 0-55.
Procedural learning | Day 0
  Assessment thanks to an experimental serial reaction task, specifically adapted for children (Gabriel et al., 2011). This is a computerized task in which are collected reaction times of children according to the spatial input occurrences on the screen, which follow a fixed procedure that is to be implicit learned (procedural learning).

SECONDARY OUTCOMES:
DNA sampling | Day 0
  The complete sequencing of FoXP2 gene, as well as the genotyping of the 44 single nucleotide polymorphisms (SNPs), located in the risk haplotypes identified in ATP2C2 (Newbury et al., 2009), CMIP (Newbury et al., 2009), CNTNAP2 (Vernes et al. 2008) genes and in the KIAA0319/TTRAP/THEM2 locus (Pinel et al., 2012), will be conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France